CLINICAL TRIAL: NCT04922554
Title: A Ph. 2, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy, Safety, & Tolerability of Oral Omadacycline in Adults With NTM Pulmonary Disease Caused by Mycobacterium Abscessus Complex
Brief Title: Oral Omadacycline vs. Placebo in Adults With NTM Pulmonary Disease Caused by Mycobacterium Abscessus Complex (MABc)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTK0796-NTM-20203
Record Dates: First submitted 2021-05-18; First posted 2021-06-10 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mycobacterium Infections, Nontuberculous; Mycobacterium Abscessus Infection; Nontuberculous Mycobacterial Lung Disease; Nontuberculous Mycobacterial Pulmonary Infection
Keywords: Nontuberculous Mycobacteria (NTM); Mycobacterium abscessus complex (MABc); NTM pulmonary disease; NTM lung disease
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — omadacycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omadacycline 300 mg PO (Experimental): omadacycline 150 mg tablets (x 2) administered orally, once daily, q24h
  Interventions: Drug: Omadacycline Oral Tablet
- Placebo PO (Placebo Comparator): Placebo tablets resembling omadacycline (x 2) administered once daily, q24h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omadacycline Oral Tablet — omadacycline 300 mg orally, once daily (150 mg tablets x 2)
  Other Names: Nuzyra
  Arms: Omadacycline 300 mg PO
Drug: Placebo — placebo tablets resembling omadacycline orally, once daily (x 2 tablets)
  Other Names: placebo tablets
  Arms: Placebo PO

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of oral omadacycline as compared to placebo in the treatment of adults with Nontuberculous Mycobacterial (NTM) pulmonary disease caused by Mycobacterium abscessus complex (MABc)

DETAILED DESCRIPTION:
The total duration of subject participation in the study is approximately 5 months which includes a total duration of study treatment for approximately 3 months (84 days). Eligible participants will be randomized 1.5:1 to receive 3 months of treatment with either omadacycline or placebo (monotherapy). The study will use a double-dummy design in order to maintain the study blinding.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a diagnosis of Nontuberculous Mycobacterial pulmonary disease caused by MABc
* Has at least 2 of the following NTM-infection symptoms present at Screening and Baseline: chronic cough, coughing up blood (hemoptysis), wheezing, chest pain, frequent throat clearing, phlegm or sputum production, shortness of breath, fatigue, fever, night sweats, poor appetite, and/or weight loss.
* At least 1 positive pulmonary (sputum) culture for MABc in the 6 months prior to Screening and 1 positive culture at Screening
* Radiographic evidence of MABc infection via computed tomography (CT) scan of the chest within 3 months prior to Screening
* In the opinion of the investigator, guideline-directed antibiotic therapy for treatment of MABc will not be required within the next 3 months, and a delay, in order for the subject to participate in a placebo-controlled clinical trial, is considered reasonable and clinically acceptable
* Additional inclusion criteria as per protocol

Key Exclusion Criteria:

* Has received antibiotic treatment within 6 months prior to Screening for MABc or MAC
* Has received systemic or inhaled antibiotic therapy (other than chronic macrolide therapy) within 4 weeks prior to Screening
* Has any of the following medical conditions:
* Active pulmonary malignancy, or any type of malignancy requiring chemotherapy or radiation within 1 year prior to Screening
* Active allergic bronchopulmonary mycosis, or any other condition requiring chronic treatment with systemic corticosteroids within 90 days prior to Screening
* Radiologic evidence of cavitary disease
* Known active pulmonary tuberculosis
* Cystic fibrosis
* History of lung transplantation
* Another advanced lung disease with a known percent predicted forced expiratory volume in 1 second < 30%.
* Disseminated or extra-pulmonary NTM disease
* Has been previously treated with omadacycline
* Has a history of hypersensitivity or allergic reaction to tetracyclines
* Additional exclusion criteria as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Chair — Paratek Pharmaceuticals Inc
Locations (17):
- United States (17):
  - Stanford University, Stanford, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Infectious Disease Consultants of the Treasure Coast, Vero Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Louisiana State University Medical Center Health Sciences Center-New Orleans Section of Pulmonary/Critical Care & Allergy/Immunology, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health, New Hyde Park, New York
  - Einstein/Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jahanbakhsh S, Howland J, Ndayishimiye Uwineza MO, Thwaites MT, Pillar CM, Serio AW, Anastasiou DM, Hufnagel DA. Evaluation of omadacycline against intracellular Mycobacterium abscessus in an infection model in human macrophages. JAC Antimicrob Resist. 2023 Sep 15;5(5):dlad104. doi: 10.1093/jacamr/dlad104. eCollection 2023 Oct. PMID 37720564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, double-blind, placebo-controlled study evaluating the efficacy and safety of omadacycline in adult participants with nontuberculous mycobacterial pulmonary disease caused by Mycobacterium abscessus complex.
Pre-assignment Details: A total of 66 participants were enrolled at 17 sites in the US.
Groups:
- Omadacycline 300 mg: Participants received omadacycline 300 mg orally (PO) (administered as two 150 mg tablets) every 24 hours (q24h).
- Placebo: Participants received matching placebo PO (administered as two tablets) q24h.
Period: Overall Study
Arm/Group | Omadacycline 300 mg | Placebo
Started | 41 | 25
Completed | 36 | 25
Not Completed | 5 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of test article.
Groups:
- Omadacycline 300 mg: Participants received omadacycline 300 mg PO (administered as two 150 mg tablets) q24h.
- Total: Total of all reporting groups
Arm/Group | Omadacycline 300 mg | Placebo | Total
Number analyzed (Participants) | 41 | 25 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (9.61) | 72.8 (7.64) | 70.6 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 15 | 45
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 36 | 23 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response on NTM Symptom Assessment Scale at Day 84
Description: A clinical responder is defined as a participant who shows improvement in at least 50% of baseline symptoms on the NTM Symptom Assessment Questionnaire at the Day 84 Visit. This self-administered tool assesses 12 common NTM symptoms, each rated on a 4-point scale (absent, mild, moderate, severe), reflecting the participant's overall impression over the past week. The questionnaire is completed solely by the participant, without any interpretation from clinicians or site staff.
Time Frame: Day 1 to Day 84
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Percentage of participants | 34.1 | 20.0
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — Endpoints are summarized using descriptive statistics. Inferential testing of pre-specified hypothesis was not completed; p = 0.2182, Chi-squared — Nominal p-values are provided for descriptive purposes; Analysis stratified by prior NTM antibiotic treatment was not performed due to small sample size in one randomization stratification subgroup; Difference in response rates = 14.15

2. Primary Outcome: Percentage of Participants With Clinical Response on NTM Symptom Assessment Scale at Day 84 With no Deterioration in Severity of Symptoms That Were Present at Baseline.
Description: A clinical responder is defined as a participant who shows improvement in at least 50% of baseline symptoms with no deterioration of symptoms present at baseline on the NTM Symptom Assessment Questionnaire at the Day 84 Visit. This self-administered tool assesses 12 common NTM symptoms, each rated on a 4-point scale (absent, mild, moderate, severe), reflecting the participant's overall impression over the past week. The questionnaire is completed solely by the participant, without any interpretation from clinicians or site staff.
Time Frame: Day 1 to Day 84
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
percentage of participants | 34.1 | 12.0
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0460, Chi-squared — Nominal p-values are provided for descriptive purposes; [statistical method as in outcome 1, analysis 1]; Difference in response rates = 22.15

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE is an adverse event that occurred on or after first dose of test article and those existing AEs that worsened on or after first dose of test article. An SAE is an adverse event that results in death, is life-threatening, requires hospitalization or extends an existing one, causes significant or lasting disability/incapacity, or leads to a congenital anomaly or birth defect. Additionally, events that may not meet these criteria but are medically significant can also be classified as SAEs.
Time Frame: From screening period (up to 8 weeks prior to randomization) through Day 114 (at any study timepoint)
Population: Safety Analysis Set included all participants who received at least 1 dose of test article.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants
  TEAEs | 35 | 21
  SAEs | 0 | 2

4. Primary Outcome: Change From Baseline in Laboratory Test Parameters - Hepatic and Enzymatic Biomarkers
Description: To assess the incidents of abnormal hepatic and enzymatic biomarkers following 84 days of IP administration
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Units per litre
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Units per litre
  Alkaline Phosphatase: number analyzed (Participants) | 39 | 25
  Alkaline Phosphatase | -3.3 (14.46) | -3.0 (11.22)
  Alanine Aminotransferase: number analyzed (Participants) | 39 | 25
  Alanine Aminotransferase | 10.4 (17.19) | -1.4 (9.74)
  Aspartate Aminotransferase: number analyzed (Participants) | 39 | 25
  Aspartate Aminotransferase | 3.9 (8.72) | -3.0 (11.88)
  Creatine Kinase: number analyzed (Participants) | 39 | 25
  Creatine Kinase | 2.5 (28.76) | -26.6 (116.68)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 39 | 25
  Gamma Glutamyl Transferase | 1.7 (14.35) | -0.6 (12.83)
  Lipase: number analyzed (Participants) | 39 | 25
  Lipase | 3.5 (16.50) | -2.2 (8.39)

5. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Laboratory Parameter
Description: Laboratory PCS event is defined as at least a 2 grade increase from baseline based on the Division of Microbiology and Infectious Diseases (DMID) v5.0.
Time Frame: Day 1 through Day 84 (at any study timepoint)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants
  Alkaline Phosphatase | 0 | 0
  Alanine Aminotransferase | 2 | 0
  Aspartate Aminotransferase | 0 | 0
  Calcium | 0 | 0
  Creatinine | 0 | 0
  Gamma Glutamyl Transferase | 0 | 0
  Lipase | 3 | 0
  Magnesium | 0 | 0
  Phosphate | 0 | 0
  Potassium | 0 | 0
  Sodium | 1 | 0
  Bilirubin | 0 | 0
  Neutrophils | 0 | 0
  Hemoglobin | 0 | 0
  Platelets | 0 | 0
  Leukocytes | 0 | 1

6. Primary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: To assess the incidents of abnormal blood pressure assessments following 84 days of IP administration
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Millimeter of mercury
  Systolic Blood Pressure | 4.3 (12.53) | 2.4 (12.62)
  Diastolic Blood Pressure | -0.5 (8.63) | 0.7 (10.45)

7. Primary Outcome: Change From Baseline in Heart Rate
Description: To assess the incidents of abnormal heart rate following 84 days of IP administration
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Beats per minute | 1.1 (8.66) | 0.2 (10.09)

8. Primary Outcome: Number of Participants With PCS Threshold Vital Signs Measurement
Description: To assess the incidents of PCS heart rate and blood pressure following 84 days of IP administration
Time Frame: Day 1 through Day 84 (at any study timepoint)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants
  Heart rate: >120 and increase of >=15 bpm | 0 | 0
  Heart rate: <=50 and decrease of >=15 bpm | 0 | 0
  Systolic blood pressure: >=180 and increase of >=20 mmHg | 0 | 0
  Systolic blood pressure: <=90 and decrease of >=20 mmHg | 0 | 0
  Diastolic blood pressure: >=105 and increase of >=15 mmHg | 0 | 0
  Diastolic blood pressure: <=50 and decrease of >=15 mmHg | 2 | 0
  Temperature: >38.0 | 0 | 0
  Temperature: <36.0 | 4 | 0

9. Primary Outcome: Change From Baseline in ECG PR Interval, QRS Duration, QT Interval, and QTcF Interval
Description: To assess the incidents of cardiac rhythm, PR interval, QRS interval, QT interval and QTc interval assessments following 84 days of IP administration
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
milliseconds
  PR Interval: number analyzed (Participants) | 38 | 25
  PR Interval | 9.7 (57.23) | 5.8 (40.93)
  QRS Duration: number analyzed (Participants) | 40 | 25
  QRS Duration | -0.5 (9.23) | -2.3 (5.11)
  QT Interval: number analyzed (Participants) | 40 | 25
  QT Interval | -11.7 (18.66) | -2.0 (29.63)
  QTcF Interval: number analyzed (Participants) | 40 | 25
  QTcF Interval | -8.5 (34.04) | -7.3 (68.65)

10. Primary Outcome: Number of Participants With PCS QTcF Value
Description: To assess the incidents of PCS and QTc interval assessments following 84 days of IP administration
Time Frame: Day 1 through Day 84/EOT (at any study timepoint)
Population: Safety Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 40 | 25
Participants
  > 450 msec | 3 | 5
  > 480 msec | 1 | 2
  > 500 msec | 1 | 0

11. Secondary Outcome: Change From Baseline in the Total Score of the Quality of Life - Bronchiectasis (QOL-B) Questionnaire - Emotional Functioning Domain
Description: The QOL-B is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for participants with non-cystic fibrosis bronchiectasis using a series of 37 questions. The QOL-B includes domains for physical functioning, role functioning, vitality, emotional functioning, social functioning, treatment burden, health perceptions and respiratory symptoms. For each domain, scores will be standardized on a 0 to 100 scale and higher scores represent better outcomes.
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 24
Score on a scale | 3.5 (2.05) | 2.7 (2.69)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8240, ANCOVA — ANCOVA analyzed change from baseline using treatment, prior antibiotic use, and baseline score as factors. LS mean difference = Omadacycline minus Placebo; Least square mean difference = 0.8, 95% CI 2-sided [-6.01 to 7.52]

12. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Health Perceptions Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 23
Score on a scale | 4.2 (2.43) | -0.9 (3.25)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2149, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 5.1, 95% CI 2-sided [-3.03 to 13.20]

13. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Physical Functioning Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 24
Score on a scale | 5.6 (3.21) | -2.7 (4.20)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1230, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 8.3, 95% CI 2-sided [-2.31 to 18.88]

14. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Respiratory Symptoms Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 24
Score on a scale | 7.5 (2.10) | 2.0 (2.75)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1168, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 5.5, 95% CI 2-sided [-1.41 to 12.43]

15. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Role Functioning Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 23
Score on a scale | 7.4 (2.14) | 0.9 (2.86)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0743, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 6.5, 95% CI 2-sided [-0.66 to 13.66]

16. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Social Functioning Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 23
Score on a scale | 9.6 (2.45) | 2.6 (3.27)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0899, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 7.1, 95% CI 2-sided [-1.13 to 15.23]

17. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Treatment Burden Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 27 | 15
Score on a scale | 2.8 (2.38) | 2.3 (3.20)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.9019, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 0.5, 95% CI 2-sided [-7.60 to 8.59]

18. Secondary Outcome: Change From Baseline in the Total Score of the QOL-B Questionnaire - Vitality Domain
Description: as for outcome 11
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT analysis set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 24
Score on a scale | 9.3 (2.50) | -4.3 (3.27)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0015, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 13.7, 95% CI 2-sided [5.43 to 21.89]

19. Secondary Outcome: Change From Baseline in Global Score and Individual Domain Scores of the SGRQ - Total Score
Description: The SGRQ is a disease-specific, 50-item instrument designed to measure the impact of obstructive airways disease on overall health, daily life, and perceived well-being in participants. It consists of three domains: Symptoms (distress from respiratory symptoms), Activity (limitations in mobility and physical activity), and Impacts (effects on employment, self-management, and medication needs). Scores range from 0 (no impairment) to 100 (maximum impairment) for each domain. The SGRQ Total Score is calculated by dividing the total score values of all positive responses across all domains in the questionnaire by the maximum possible total score that a participant could have achieved, and then multiplying the result by 100. Higher scores indicate worse health status
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Score on a scale
  Activity score | -2.7 (2.50) | -3.6 (3.17)
  Impact score | -3.7 (2.29) | -3.5 (2.99)
  Symptom score | -5.6 (2.43) | -0.6 (3.11)
  Total score | -3.7 (2.06) | -3.0 (2.67)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8269, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = 0.9, 95% CI 2-sided [-7.26 to 9.05] — Treatment comparison of Omadacycline and Placebo for activity score has been presented
Statistical Analysis 2: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.9584, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = -0.2, 95% CI 2-sided [-7.74 to 7.35] — Treatment comparison between Omadacycline and Placebo for impact score has been presented
Statistical Analysis 3: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2123, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = -5.0, 95% CI 2-sided [-12.88 to 2.92] — Treatment comparison between Omadacycline and Placebo for symptom score has been presented
Statistical Analysis 4: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.8161, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = -0.8, 95% CI 2-sided [-7.58 to 5.99] — Treatment comparison between Omadacycline and Placebo for total score has been presented

20. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System Short Form v1.0 - Fatigue 7a Daily (PROMIS-7a) Score
Description: The PROMIS Fatigue is a self-administered questionnaire that assesses fatigue and its impact on physical, mental, and social activities. The fatigue short form is universal rather than disease-specific and assesses fatigue over the past 7 days. Participants respond to each of the 7 items using a 5-point Likert scale (e.g., "Not at all" to "Very much") and item responses are summed to produce a raw total score. Raw scores are converted to T-scores using standardized PROMIS scoring tables. The average change in PROMIS Fatigue T-scores was calculated for each study arm. The PROMIS Fatigue T-score is a standardized score (mean = 50, SD = 10) where higher scores indicate greater fatigue severity. A negative change from baseline (i.e., lower T-scores over time) indicates improvement in fatigue symptoms, whereas a positive change (i.e., higher T-scores) indicates worsening of fatigue.
Time Frame: Day 1 (Baseline) to Day 84/EOT
Population: ITT Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 40 | 24
score on a scale | -4.3 (1.01) | 1.3 (1.30)
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0010, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Least square mean difference = -5.7, 95% CI 2-sided [-8.95 to -2.38]

21. Secondary Outcome: Number of Participants With Improvement in Patient Clinical Impression of Change (PGI-C)
Description: The PGI-C is a self-administered, single question assessed using a 7-point scale that measures a participant's perceived change in clinical status and overall improvement. Participants with improvement includes: Very much improved, much improved, minimally improved; participants without improvement include: no change, minimally worse, much worse, very much worse.
Time Frame: Day 1 to Day 84/EOT
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants | 31 | 9
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0020, Fisher Exact; Difference in improvement rates = 39.61, 95% CI 2-sided [16.66 to 62.56]

22. Secondary Outcome: Number of Participants Reporting "Not Present or Mild Severity" in Patient Clinical Impression of Severity (PGI-S)
Description: The PGI-S is a self-administered, single question assessed using a 7-point scale that measures a participant's perception of disease severity. Participants with severity Not present or Mild include: not present, very mild, mild; Participants with severity Moderate or Severe include: moderate, moderately severe, severe, extremely severe.
Time Frame: Day 84/EOT
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants | 26 | 12
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3051, Fisher Exact; Difference in improvement rates = 15.41, 95% CI 2-sided [-9.10 to 39.93]

23. Secondary Outcome: Number of Participants With Clinical Global Impression - Severity of Illness (CGI-S)
Description: The CGI-S is administered by an experienced clinician who is familiar with the disease under study. The CGI-S is a 1-item observer-rated scale that rates illness severity based upon observed and reported symptoms, behavior, and function over the past seven days.
Time Frame: Day 84/EOT
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants
  Normal, not at all ill | 14 | 4
  Borderline ill | 9 | 8
  Mildly ill | 11 | 9
  Moderately ill | 6 | 4
  Markedly ill | 0 | 0
  Severely ill | 1 | 0
  Among the most extremely ill participants | 0 | 0
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3552, Wilcoxon rank sum test

24. Secondary Outcome: Number of Participants With Clinical Global Impression - Improvement (CGI-I)
Description: The CGI-I is a single-item, observer-rated measure using a 7-point scale to assess overall improvement in a participant's condition due to drug treatment. Participants with improvement includes: very much improved, much improved, minimally improved; participants without improvement include: no change, minimally worse, much worse, very much worse.
Time Frame: Day 1 to Day 84/EOT
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants | 29 | 11
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0753, Wilcoxon rank sum test

25. Secondary Outcome: Number of Participants With New Symptoms With a Severity Worse Than Mild on the NTM Symptom Assessment Questionnaire at Any Time Post-baseline
Description: The NTM symptom assessment questionnaire is a self-administered tool which assesses 12 common NTM symptoms on a 4-point scale (absent, mild, moderate, severe), reflecting the participant's overall impression over the past week. The questionnaire is completed solely by the participant, without any interpretation from clinicians or site staff.
Time Frame: Day 1 through Day 84 (at any study timepoint)
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Participants | 4 | 6

26. Secondary Outcome: Number of Participants With Decreased Semi-Quantitative Score of Mycobacterial Sputum Culture From Day 1 to Day 84
Description: Semi-quantitative score is derived based on growth in liquid medium, growth on agar plate, and colony count on agar plate; the score ranges from 0 to 6. A reduction in the semi-quantitative score reflects a decrease in the quantitative mycobacterial load.
Time Frame: Day 1 to Day 84
Population: ITT Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 34 | 24
Participants | 26 | 11
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0168, Chi-squared; Odds Ratio (OR) = 3.84, 95% CI 2-sided [1.24 to 11.87]

27. Secondary Outcome: Time to Growth in Liquid Medium Only
Description: Time to growth in liquid medium only is defined as the number of days from the date of study drug administration to the date of the first assessment where growth is detected in liquid medium only. The analysis was based on Kaplan Meier Estimation for Growth in Liquid Medium Only (Day). If there is no culture result indicating growth in liquid medium only and the culture plates are negative, the date of the first negative culture is used for determination of time to growth in liquid medium only.
Time Frame: Day 1 through Day 84 (at any study timepoint)
Population: ITT Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 37 | 23
Days | 34 [28 to 83] | NA [28 to NA] — Not Applicable (NA) indicates median and upper limit of CI was not calculated due to less than 50% of participants had growth in liquid medium only.
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0233, Log Rank

28. Secondary Outcome: Time to First Negative Sputum Culture
Description: Time to first negative sputum culture is defined as the number of days from the date of study drug administration to the date of the first negative sputum culture. The analysis was based on Kaplan Meier Estimation for Negative Sputum Culture (Day).
Time Frame: Day 1 through Day 84 (at any study timepoint)
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Omadacycline 300 mg | Placebo
Number analyzed (Participants) | 41 | 25
Days | 30 [28 to 84] | NA [30 to NA] — NA indicates median and upper limit of CI was not calculated due to less than 50% of participants had growth in liquid medium only.
Statistical Analysis 1: Comparison: Omadacycline 300 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0349, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from screening period (up to 8 weeks prior to randomization) through the final Follow-up assessment, which occurred up to 30 days after the last dose of study treatment, with the treatment period lasting for 84 days.
Arm/Group | Omadacycline 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/25
Other Adverse Events (participants affected / at risk) | 35/41 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omadacycline 300 mg (N=41) | Placebo (N=25)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omadacycline 300 mg (N=41) | Placebo (N=25)
Nausea (Gastrointestinal disorders) | 22 (37) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (15) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 7 (8) | 4 (5)
Fatigue (General disorders) | 7 (8) | 1 (1)
Vessel puncture site reaction (General disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04922554/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT04922554/SAP_001.pdf